CLINICAL TRIAL: NCT00124449
Title: A Phase II Study of Abatacept Versus Placebo to Assess the Prevention of Rheumatoid Arthritis (RA) in Adult Patients With Undifferentiated Arthritis Who Are at High Risk for the Development of RA
Brief Title: Study of Abatacept Versus Placebo to Assess the Prevention of Rheumatoid Arthritis (RA) in Adult Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: IM101-046
Record Dates: First submitted 2005-06-30; First posted 2005-07-28 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Abatacept
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Abatacept — solution, intravenous injection, monthly, 169 days
  weight based:
  <60 kg = 500 mg
  60 to 100 kg = 750 mg
  >100 kg = 1 g
  Other Names: Orencia
  Arms: 1
Drug: placebo — solution, intravenous injection, 0 mg, monthly, 169 days
  Arms: 2

SUMMARY:
The purpose of this study is to assess if Abatacept given for six months will prevent rheumatoid arthritis (RA) in patients who are at risk for the development of RA in comparison to placebo. High risk patients are defined as those having a positive laboratory test for anti-cyclic citrullinated peptide (anti-CCP2).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of undifferentiated arthritis
* Clinical synovitis of two or more joints
* At least one but not more than three of the criteria for diagnosis of RA (1987).
* No prior disease modifying anti-rheumatic drugs (DMARDs)/biologics.
* Duration of disease must be 18 months or less.
* Positive for antibodies against cyclic citrullinated peptides.

Exclusion Criteria:

* Women of child bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy.
* Active vasculitis of a major organ system.
* Severe or recurrent bacterial infection.
* History of cancer in the last five years except certain skin cancers.
* Herpes zoster that resolved less than 2 months prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-02; Primary Completion 2007-05 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (48):
- United States (20):
  - Local Institution, Huntsville, Alabama
  - Local Institution, Mobile, Alabama
  - Local Institution, Huntington Beach, California
  - Local Institution, Los Angeles, California
  - Local Institution, Boulder, Colorado
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Chicago, Illinois
  - Local Institution, Evansville, Indiana
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Cumberland, Maryland
  - Local Institution, Hagerstown, Maryland
  - Local Institution, Duluth, Minnesota
  - Local Institution, Durham, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Willow Grove, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Austin, Texas
  - Local Institution, Arlington, Virginia
- Australia (4):
  - Local Institution, Cairns, Queensland
  - Local Institution, Clayton, Victoria
  - Local Institution, Malvern, Victoria
  - Local Institution, Shenton Park, Western Australia
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Leuven
- France (2):
  - Local Institution, Paris
  - Local Institution, Strasbourg
- Germany (5):
  - Local Institution, Berlin
  - Local Institution, Dresden
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Heidelberg
- Italy (3):
  - Local Institution, Bari
  - Local Institution, Ferrara
  - Local Institution, Milan
- Mexico (4):
  - Local Institution, León, Guanajuato
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Guadalajara, Mexico City
  - Local Institution, Morelia, Michioacan
- Local Institution, Ponce, Puerto Rico
- Spain (5):
  - Local Institution, A Coruña
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Oviedo
  - Local Institution, Seville
- United Kingdom (2):
  - Local Institution, Liverpool, Merseyside
  - Local Institution, Leeds, North Yorkshire

REFERENCES:
- [Background] Emery P, Durez P, Dougados M, Legerton CW, Becker JC, Vratsanos G, Genant HK, Peterfy C, Mitra P, Overfield S, Qi K, Westhovens R. Impact of T-cell costimulation modulation in patients with undifferentiated inflammatory arthritis or very early rheumatoid arthritis: a clinical and imaging study of abatacept (the ADJUST trial). Ann Rheum Dis. 2010 Mar;69(3):510-6. doi: 10.1136/ard.2009.119016. Epub 2009 Nov 23. PMID 19933744

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 184 participants were screened, 127 were enrolled but not randomized (5 withdrew consent; 120 no longer met study criteria; 2 other reasons). 57 participants were randomized, 1 participant was randomized but not treated.
Groups:
- Abatacept: Abatacept by intravenous (IV) infusion, dose based on participant's body weight at the screening visit
- Placebo: Placebo (dextrose 5% in water [D5W] or normal saline [NS]) by IV infusion.
Period: 6-month Double-Blind Treatment Period
Arm/Group | Abatacept | Placebo
Started | 28 | 28
Completed | 22 | 17
Not Completed | 6 | 11
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 3 | 8
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Poor/Noncompliance | 1 | 0
Not completed — Sponsor request | 0 | 1
Not completed — Exposure to mycobacterium tuberculosis | 0 | 1
Period: 18-Month Untreated Observation Period
Arm/Group | Abatacept | Placebo
Started | 22 | 17
Completed Year 1 of Study | 14 | 9
Completed | 7 | 4
Not Completed | 15 | 13
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 11 | 12
Not completed — Lost to Follow-up | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Poor/Noncompliance | 1 | 0
Not completed — Relocated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Abatacept: Abatacept by IV infusion, dose based on participant's body weight at the screening visit
- Total: Total of all reporting groups
Arm/Group | Abatacept | Placebo | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (10.9) | 44.7 (12.1) | 44.8 (11.4)
Age, Continuous [Median (Full Range); unit: years] | 43.5 [23.0 to 74.0] | 44.0 [26.0 to 71.0] | 44.0 [23.0 to 74.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 25 | 23 | 48
  Black | 1 | 3 | 4
  Asian | 1 | 1 | 2
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  North America | 6 | 5 | 11
  South America | 5 | 2 | 7
  Europe | 17 | 21 | 38
Months of Undifferentiated Inflammatory Arthritis (UA) [Mean (Standard Deviation); unit: Months] | 8.8 (4.2) | 7.1 (4.4) | 7.9 (4.3)
Weight [Mean (Standard Deviation); unit: Kilograms] | 75.9 (22.5) | 70.9 (13.9) | 73.4 (18.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Diagnosis of Rheumatoid Arthritis (RA) by American Rheumatism Association (ARA) Criteria and/or Discontinued Due to Lack of Efficacy
Description: ARA criteria is a 7-item tool for RA classification purposes; a patient is said to have RA (meeting endpoint) if he or she has satisfied at least 4 of the 7 criteria. If a participant discontinued due to lack of efficacy, he/she was regarded as meeting primary endpoint also.
Time Frame: 12 months
Population: Randomized and treated participants were included in analysis if they were RA positive and/or were discontinued due to lack of efficacy. (Those who discontinued due to reasons other than lack of efficacy in 1-year window were excluded from the analysis). 1 participant in Placebo group was excluded due to presence of RA at baseline.
Measure: Number; unit: Participants
Groups:
- Abatacept: Abatacept by intravenous (IV) infusion, dose based on subject's body weight at the screening visit
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 26 | 24
Participants | 12 | 16

2. Secondary Outcome: Number of Participants With a Diagnosis of RA by 1987 ARA Criteria and/or Discontinued Due to Lack of Efficacy
Description: ARA criteria is a 7-item tool for classification purposes; a patient is said to have RA (meeting endpoint) if he or she has satisfied at least 4 of the 7 criteria. If a participant discontinued due to lack of efficacy, he/she was regarded as meeting endpoint also.
Time Frame: 24 months
Population: Randomized and treated participants were included in analysis if they were RA positive and/or were discontinued due to lack of efficacy. (Those who discontinued due to reasons other than lack of efficacy in 2-year window were excluded from the analysis). 1 subject in the Placebo group is excluded due to presence of RA at baseline.
Measure: Number; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 23 | 24
Participants | 17 | 21

3. Secondary Outcome: Number of Participants With Undifferentiated Inflammatory Arthritis (UA) Who Develop Another Rheumatic Disease
Description: Clinical diagnosis of other rheumatic diseases at 12 and 24 months. If a participant discontinued due to lack of efficacy, he/she was regarded as meeting endpoint also.
Time Frame: 12 months, 24 months
Population: n=Randomized and treated participants who were RA positive and/or were discontinued due to lack of efficacy. (Those who discontinued due to reasons other than lack of efficacy in the 1- or 2-year window were excluded from the analysis).1 participant in Placebo group was excluded due to the presence of RA at baseline.
Measure: Number; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
Participants
  12 months (n=26; n=24) | 0 | 0
  24 months (n=23; n=24) | 0 | 0

4. Secondary Outcome: Change From Baseline in Radiographic Erosion and Joint Space Narrowing Score at 6 Months, 12 Months, and 24 Months
Description: Mean change from baseline using the Genant-Modified Sharp Score. Erosion score=assessment of 14 sites in each hand and wrist + 6 joints in each foot, using an 8-point scale from 0 (no erosions) to 3.5 (erosions of 100% or articular surfaces). Joint score= assessment of 13 sites in each wrist and hand + 6 sites in each foot using a 9-point scale from 0 (normal) to 4.0 (definite ankylosis). As-observed data. Change from Baseline=postbaseline score at timepoint (6 or 12 or 24 months) minus baseline score; a lower value signifies improvement.
Time Frame: Baseline, 6 months, 12 months, 24 months
Population: n=participants with a score at baseline and at timepoint
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale
  Erosion Score 6 months (n=22; n=21) | 0.13 (0.09) | 0.46 (0.24)
  Joint Space Narrowing 6 months (n=22; n=21) | 0.00 (0.00) | 0.01 (0.01)
  Total Score 6 months (n=22; n=21) | 0.13 (0.09) | 0.47 (0.24)
  Erosion Score 12 months (n=17; n=11) | 0.02 (0.04) | 0.85 (0.39)
  Joint Space Narrowing 12 months (n=17; n=11) | 0.00 (0.00) | 0.26 (0.22)
  Total Score 12 months (n=17; n=11) | 0.02 (0.04) | 1.11 (0.56)
  Erosion Score 24 months (n=7; n=3) | 0.04 (0.04) | -0.17 (0.17)
  Joint Space Narrowing 24 months (n=7; n=3) | 0.00 (0.00) | 0.00 (0.00)
  Total Score 24 months (n=7; n=3) | 0.04 (0.04) | -0.17 (0.17)

5. Secondary Outcome: Change From Baseline in Total Erosion, Edema, Synovitis Scores at 6 Months, 12 Months, and 24 Months
Description: Mean change from baseline. Degree of synovitis and structural joint damage (erosion, edema) of the carpal and metacarpophalangeal joints, as measured by magnetic resonance imaging (MRI) scores using the European League Against Rheumatism (EULAR)-Outcome Measures in Rheumatology Clinical Trials (OMERACT) assessment. Edema scale=0 (no bone involved) to 3 (67% to 100% of bone involved). Synovitis scale=0 (normal) and 1-3 (mild, moderate, severe. Bone erosion scale=0 (0% of bone involved) to 10 (91% to 100% of bone involved). Change from baseline=postbaseline score at timepoint - baseline score.
Time Frame: Baseline, 6 months, 12 months, 24 months
Population: All randomized and treated participants (n=number of participants with baseline and postbaseline measurements). MRIs were done only in participants at European Union sites.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale
  Erosion Score at 6 months (n=11; n=10) | 0.45 (0.37) | 1.20 (1.09)
  Edema Score at 6 months (n=11; n=10) | -1.64 (1.48) | 1.40 (1.59)
  Synovitis Score at 6 months (n=11; n=10) | 0.27 (0.56) | 1.60 (1.23)
  Erosion Score at 12 months (n=9; n=6) | 0.00 (0.17) | 5.00 (3.20)
  Edema Score at 12 months (n=9; n=6) | 0.22 (0.49) | 6.67 (4.22)
  Synovitis Score at 12 months (n=9; n=6) | 0.22 (0.22) | 2.33 (1.61)
  Erosion Score at 24 months (n=5; n=2) | 0.80 (0.49) | 0.00 (0.00)
  Edema Score at 24 months (n=5; n=2) | 0.20 (0.20) | 0.50 (0.50)
  Synovitis Score at 24 months (n=5; n=2) | 0.60 (0.60) | 1.50 (2.50)

6. Secondary Outcome: Number of Participants With Persistent Symptomatic Clinical Synovitis
Description: Synovitis, assessed by clinical signs and symptoms
Time Frame: 6, 12, and 24 months
Population: All randomized and treated participants (n=number of participants with assessment at baseline and timepoint)
Measure: Number; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
Participants
  6 months (n=5; n=12) | 4 | 12
  12 months (n=11; n=7) | 10 | 7
  24 months (n=3; n=2) | 3 | 2

7. Secondary Outcome: Short Form-36 (SF-36) Physical and Mental Component Summary (PCS and MCS) Scores - Mean Change From Baseline
Description: SF-36, a 36-item instrument that covers 8 quality of life domains, which were used to derive the physical and mental component summary scores, which ranged from 0 to 100, with higher scores indicating a better quality of life. Change from baseline=postbaseline - baseline value; a higher value signifies improvement.
Time Frame: 6 months, 12 months, 24 months
Population: All randomized and treated participants (n=number of participants with baseline and postbaseline measurements)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale
  PCS, 6 months (n=26; n=20) | 10.23 (1.68) | 1.95 (1.52)
  MCS, 6 months (n=26; n=20) | 2.54 (1.33) | -0.30 (1.29)
  PCS, 12 months (n=20; n=14) | 3.83 (2.38) | -0.81 (2.26)
  MCS, 12 months (n=20; n=14) | 2.50 (1.75) | -2.89 (2.85)
  PCS, 24 months (n=7; n=5) | 2.46 (3.15) | -2.17 (6.44)
  MCS, 24 months (n=7; n=5) | 3.75 (1.99) | -3.30 (7.58)

8. Secondary Outcome: Change From Baseline in Cytokine Levels and Second Generation Anti-cyclic Citrullinated Peptide (Anti-CCP2) Antibodies at 6 Months, 12 Months, and 24 Months
Description: To assess pharmacodynamic effect of abatacept on serum levels of autoantibodies, mean change from baseline in cytokines (interleukin-6 [IL-6], interleukin-1B [IL-1B], tumor necrosis factor Alpha [TNF-Alpha], Matrix Metalloproteinase 3T [MMP3T], and anti-CCP2), as measured by standard laboratory investigations, were assessed. Change from baseline=postbaseline value at timepoint (6 or 12 or 24 months) minus baseline value; a lower value signifies improvement.
Time Frame: Baseline, 6 Months, 12 months, 24 months
Population: All randomized and treated participants (n=number of participants with baseline and postbaseline measurements).
Measure: Mean (Standard Error); unit: laboratory values
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
laboratory values
  IL6 at 6 months (n=19, n=18) | -4.49 (1.78) | 1.08 (0.72)
  IL6 at 12 months (n=13, n=7) | -0.14 (1.61) | 6.37 (3.81)
  IL6 at 24 months (n=5, n=3) | -3.44 (3.54) | 0.90 (1.51)
  IL1B at 6 months (n=18, n=18) | -0.12 (0.07) | -0.09 (0.08)
  IL1B at 12 months (n=13, n=7) | -0.09 (0.07) | -0.24 (0.21)
  IL1B at 24 months (n=5, n=1) | 0.20 (0.20) | 0.00 (0.00)
  TNF-Alpha at 6 months (n=18, n=18) | -1.70 (1.29) | 0.07 (0.28)
  TNF-Alpha at 12 months (n=13, n=7) | -0.50 (0.25) | -0.10 (0.33)
  TNF-Alpha at 24 months (n=13, n=7) | -0.82 (0.47) | -0.03 (0.03)
  MMP3T at 6 months (n=20, n=19) | -2.29 (4.86) | 14.34 (9.85)
  MMP3T at 12 months (n=15, n=9) | -2.55 (3.08) | 25.34 (14.59)
  MMP3T at 24 months (n=6, n=3) | 6.73 (6.93) | 3.10 (3.45)
  Anti-CCP2 antibodies at 6 months (n=21, n=19) | -94.5 (29.49) | 16.32 (21.49)
  Anti-CCP2 antibodies at 12 months (n=14, n=10) | -6.46 (48.09) | 149.5 (64.38)
  Anti-CCP2 antibodies at 24 months (n=6, n=3) | 3.43 (53.85) | -35.1 (55.65)

9. Secondary Outcome: Number of Participants With Anti-CCP2 Positive and/or Rheumatoid Factor (RF) Positive Over Time
Description: To assess the pharmacodynamic effect of abatacept on serum levels of autoantibodies, number of participants with Anti-CCP2 Positive of Rheumatoid Factor (RF) positive
Time Frame: Day 1, 6 months, 12 months, 24 months
Population: All randomized and treated participants (n=number of participants with measure at timepoint).
Measure: Number; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
Participants
  Anti-CCP2 Positive on Day 1 (n=28, n=28) | 28 | 28
  Anti-CCP2 Positive at 6 months (n=22, n=19) | 20 | 19
  Anti-CCP2 Positive at 12 months (n=15, n=10) | 13 | 10
  Anti-CCP2 Positive at 24 months (n=6, n=3) | 5 | 3
  RF on Day 1 (n=28, n=28) | 24 | 20
  RF at 6 months (n=22, n=20) | 13 | 14
  RF at 12 months (n=15, n=10) | 11 | 8
  RF at 24 months (n=6, n=3) | 3 | 3

10. Secondary Outcome: Frequency of Human Leukocyte Antigen (HLA) Typing
Description: To assess the pharmacodynamic effect of abatacept on serum levels of autoantibodies, a blood sample was obtained for HLA typing to determine the presence or absence of alleles associated with RA susceptibility and severity (shared epitope alleles HLA-DRB10401 and HLA-DRB10404).
Time Frame: Day 1
Population: All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
participants
  Missing | 4 | 7
  Undetected | 11 | 10
  Detected | 13 | 11

11. Secondary Outcome: DAS 28 C Reactive Protein (CRP) Score - Mean Change From Baseline
Description: The DAS 28 (CRP) is a composite of 4 variables: 28 tender joint count, 28 swollen joint count, CRP, and subject assessment of disease activity measure on a VAS of 100 mm. Change from Baseline=postbaseline score-baseline score; a lower value signifies improvement.
Time Frame: 6 months, 12 months, 24 months
Population: All randomized and treated participants (n=the number of participants with baseline and postbaseline measurements).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale
  6 Months (n=20; n=20) | -1.13 (0.20) | 0.01 (0.26)
  12 Months (n=18; n=13) | -0.50 (0.22) | -0.05 (0.42)
  24 Months (n=6; n=4) | -0.33 (0.33) | 0.69 (1.16)

12. Secondary Outcome: Number of Participants With a DAS 28 (CRP) Score of ≤3.2 (Low Disease Activity) or <2.6 (in Remission)
Description: The DAS 28 (CRP) is a composite of 4 variables: tender joint count, swollen joint count, CRP, and subject assessment of disease activity measure on a VAS of 100 mm. Scores for disease activity are defined as low (≤ 3.2) and in remission (< 2.6).
Time Frame: 6 months, 12 months, 24 months
Population: All randomized and treated participants (n=the number of participants with baseline and postbaseline measurements).
Measure: Number; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
Participants
  ≤3.2 at 6 months (n=21; n=20) | 17 | 9
  <2.6 at 6 months (n=21; n=20) | 15 | 7
  ≤3.2 at 12 months (n=19; n=13) | 13 | 7
  <2.6 at 12 months (n=19; n=13) | 9 | 5
  ≤3.2 at 24 months (n=7; n=4) | 5 | 2
  <2.6 at 24 months (n=7; n=4) | 4 | 2

13. Secondary Outcome: Number of Subjects With Health Assessment Questionnaire (HAQ) Disability Index Response
Description: This questionnaire includes 20 questions assessing physical function in 8 domains. The questions are evaluated on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do. Higher scores indicate greater dysfunction. HAQ response =improvement of at least 0.3 units from baseline.
Time Frame: 6 months, 12 months, 24 months
Population: All randomized and treated participants (n=the number of participants with baseline and postbaseline measurements).
Measure: Number; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
Participants
  6 Months (n=26; n=25) | 16 | 6
  12 months (n=25; n=25) | 9 | 3
  24 months (n=21; n=24) | 3 | 1

14. Secondary Outcome: Overall Safety - Adverse Events (AEs), Serious AEs, and Deaths
Description: AEs were monitored at all scheduled visits of the study drug treatment and observation periods and at the follow-up visits performed 28, 56, and 85 days after the last infusion of study medication for participants who were withdrawn prematurely
Time Frame: Throughout the treatment period (6 months)
Population: All subjects who received at least 1 dose of study medication
Measure: Number; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 28 | 28
Participants
  Deaths | 0 | 0
  SAEs | 1 | 1
  AEs | 18 | 20
  Related AEs | 14 | 10
  Discontinued due to AEs | 1 | 1

15. Secondary Outcome: Number of Participants With Positive Responses for Serum Levels of Abatacept-specific Antibodies
Description: Immunogenicity, as measured by the number of positive repsonses for serum levels of abatacept-specific antibodies measured by enzyme-linked immunosorbent assays (ELISA). Postive response for whole molecule assessment was a value of > 400 and for tip assessment was ≥25.
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 27
participants | 4

ADVERSE EVENTS:
Arm/Group | BMS-188667 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/28
Other Adverse Events (participants affected / at risk) | 16/28 | 13/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-188667 (N=28) | Placebo (N=28)
SCIATICA (Nervous system disorders) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-188667 (N=28) | Placebo (N=28)
HEADACHE (Nervous system disorders) | 3 | 2
NAUSEA (Gastrointestinal disorders) | 0 | 2
VOMITING (Gastrointestinal disorders) | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 4 | 3
CONSTIPATION (Gastrointestinal disorders) | 0 | 2
RHINITIS (Infections and infestations) | 0 | 2
SINUSITIS (Infections and infestations) | 2 | 0
PHARYNGITIS (Infections and infestations) | 2 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 3
NASOPHARYNGITIS (Infections and infestations) | 3 | 2
URINARY TRACT INFECTION (Infections and infestations) | 2 | 3
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 4
PAIN (General disorders) | 0 | 2
CHILLS (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.